CLINICAL TRIAL: NCT07009015
Title: The Effect Of Health Education Intervention Program In Improving Knowledge, Attitude, And Practice Of Oral Health Among Male Primary School Children In Al-Lith Saudi Arabia: A Clustered Randomised Control Trial
Brief Title: Impact of Oral Health Program on Al-Lith Children's KAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Mohammed Khalid Salem Alsharif, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MKSalemAlsharif
Record Dates: First submitted 2025-05-21; First posted 2025-06-06 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Dental Caries in Children
Keywords: Dental caries; Oral health status; Knowledge; Attitude; Practice
MeSH Terms: conditions — Dental Caries; Behavior

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial (RCT)
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The oral health education intervention program (Other): The intervention program aims to enhance students' oral health knowledge, attitudes, and behaviors over a one-month school term through educational and practical sessions, with its effectiveness assessed before and after the intervention using a closed-ended questionnaire.
  Interventions: Other: The oral health education intervention program
- Control group: No Intervention (No Intervention): They will have their regular curriculums and normal activity routine.

INTERVENTIONS:
Other: The oral health education intervention program — The intervention program will be designed to improve oral health knowledge, attitudes, and behaviors among students over a one-month school term, carefully scheduled to avoid disrupting regular academic activities. The program consists of initial sessions focused on building students' understanding and appreciation of oral health and healthy eating habits, followed by sessions aimed at developing practical behavioral skills. The effectiveness of the program will be evaluated at three points-before the intervention, two months after, and four months post-intervention-using a closed-ended questionnaire to assess changes in knowledge, attitudes, and practices.
  Arms: The oral health education intervention program

SUMMARY:
Dental caries remains a significant global public health issue, particularly affecting children's health, development, and well-being, with inadequate knowledge, attitudes, and practices around oral health exacerbating these impacts. To address this, a cluster randomized controlled trial will be conducted in four primary schools in Al Lith City, Saudi Arabia, targeting children aged 10 to 11 years. The intervention involves interactive, classroom-based educational sessions led by a dental care professional, supplemented by take-home materials, focusing first on enhancing knowledge and attitudes, and then on developing behavioral skills for improved oral hygiene and eating habits. Participants' knowledge, attitudes, and practices will be assessed via questionnaires before, immediately after, and six months post-intervention, with data analyzed using SPSS through descriptive statistics, chi-square tests, One Way-ANOVA, and Generalized Estimating Equations. The study expects that school-based oral health education will significantly improve children's oral health knowledge and certain hygiene behaviors, as well as positively influence eating habits and patterns.

DETAILED DESCRIPTION:
Background: Dental caries is a global public health concern and impacts children's health. Good oral health status at a young age is essential for children's development, general health, and well-being. Therefore, a lack of knowledge, attitude, and practice on oral health will affect children's development, overall health, and well-being. This study aims to evaluate a brief oral health intervention in schools by a primary dental care practitioner in improving the knowledge, practice, and attitude toward oral health care among primary school children in Al Lith City, Saudi Arabia. A cluster randomized controlled trial (CRCT) will be conducted in four schools in Al Lith City, Saudi Arabia, among children aged 10 to 11 years old. Methods: 160 children will receive classroom-based interactive educational sessions delivered by a dental care professional and receive take-home literature on oral health. The first session will focus on developing the participant's knowledge and attitude toward oral health. In contrast, the second session will cover topics on behavioural skills improvement to apply the knowledge and skills gained from the first session to improve their targeted behaviours of oral hygiene and eating habits. All children will complete a questionnaire on oral health knowledge, attitude, and practice before, immediately after, and six months following the intervention. Data will be analyzed using SPSS. Data will be presented by descriptive statistics. Chi-square test will be used to determine the association between the variables of the study. One Way-ANOVA will determine the mean differences for the selected variables. A generalized Estimating Equations (GEE) will be used to test the effect of the oral health education program on the outcomes between and within the groups. Expected Results: School-based preventative oral health education delivered by primary dental care practices can improve children's knowledge of oral health and some aspects of oral hygiene behaviour. There are significant differences will be detected in eating habits and eating patterns.

ELIGIBILITY:
Inclusion Criteria:

* Primary school male students.
* Aged 10 to 11 years old.
* Students who have at least one of their parent's consents to participate in the study.

Exclusion Criteria:

* Students who are medically ill at the time of conducting the study.
* Students that are absent while conducting the study.

Ages: 10 Years to 11 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 430 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Knowledge on oral health status | (Timepoint 1 = Baseline, Timepoint 2 = 8-weeks post intervention, Timepoint 3 = 16-weeks post intervention)
  The oral health knowledge assessment consists of eighteen multiple-choice questions scored as correct (1) or incorrect (0), categorized into four domains (dentition, dental caries, gingivitis, and oral cancer), and combined into a composite index with a total possible score ranging from 0 to 18.
Attitude on oral health status | (Timepoint 1 = Baseline, Timepoint 2 = 8-weeks post intervention, Timepoint 3 = 16-weeks post intervention)
  A 12-item, five-point Likert scale questionnaire wiil be used to assess attitudes toward maintaining oral hygiene, with five negatively worded items inversely recoded, yielding total scores ranging from 12 to 60.
Practice on oral health status | (Timepoint 1 = Baseline, Timepoint 2 = 8-weeks post intervention, Timepoint 3 = 16-weeks post intervention)
  There are 12 multiple-choice questions in this part. The correct answers will be coded as the highest score, and the wrong answers will be coded as '0'. There is a maximum score of 18 and a minimum of 0.

SECONDARY OUTCOMES:
Self efficacy | (Timepoint 1 = Baseline, Timepoint 2 = 8-weeks post intervention, Timepoint 3 = 16-weeks post intervention)
  A seven-item self-reported questionnaire will be used to assess students' self-efficacy towards oral health, with respondents rating their confidence on a 5-point Likert scale ranging from "Not confident" to "Completely confident."
Social support Appraisals | (Timepoint 1 = Baseline, Timepoint 2 = 8-weeks post intervention, Timepoint 3 = 16-weeks post intervention)
  The Social Support Appraisals Scale is a 23-item questionnaire with five response options that measures the extent to which individuals feel loved, esteemed, and involved with family, friends, and others.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Iqmer Nashriq Mohd Nazan, PhD, Study Director — Universiti Putra Malaysia
Locations (1):
- Universiti Putra Malaysia, Serdang, Selangor, Malaysia